CLINICAL TRIAL: NCT06520267
Title: Prevalence of Bacteriuria, Antibiotic Susceptibility, and Treatment Response in Patients With Symptomatic Benign Prostatic Hyperplasia: a Prospective Observational Study
Brief Title: Prevalence of Bacteriuria, Antibiotic Susceptibility, and Treatment Response in Symptomatic Benign Prostatic Hyperplasia
Acronym: BPH
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Prinicpal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: IRC/1694/019
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Bacteriuria in Symptomatic Benign Prostate Hyperplasia; Antibiotic Susceptibility in Symptomatic Benign Prostate Hyperplasia; Treatment Response to Antibiotics in Symptomatic Benign Prostate Hyperplasia
Keywords: Bacteriuria; Benign Prostate Hyperplasia; Urinary Tract Infection
MeSH Terms: conditions — Bacteriuria; Prostatic Hyperplasia; Urinary Tract Infections | interventions — Anti-Infective Agents; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Urine culture and antibiotic sensitivity tests were conducted to assess the bacteriological profile among symptomatic BPH patients.The DNA of these microorganisms can be extracted and analyzed as part of the bacterial evaluation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- symptomatic BPH: All patients with symptomatic BPH attending the Urology Out-Patient Department (OPD) of the study site were enrolled. Informed and written consent was obtained from all participants. Demographic data were recorded, and detailed histories were taken regarding the duration and symptoms of BPH and relevant past history. IPSS scoring was conducted. A thorough clinical examination, including general physical, systemic, and digital rectal examination, was performed. During the rectal examination, the prostate was checked for nodules, softness, induration, or tenderness. Urine culture and antibiotic sensitivity tests were conducted to assess the bacteriological profile.
  Interventions: Drug: Antibiotic therapy

INTERVENTIONS:
Drug: Antibiotic therapy — Urine culture and antibiotic sensitivity tests were conducted to assess the bacteriological profile. The patients were then prescribed antibiotics based on susceptibility testing for a duration of 1 week.
  Other Names: Antibiotics

SUMMARY:
The goal of this prospective observational study is to identify the common pathogens and antibiotic sensitivity pattern in urine samples of men with symptomatic BPH and to assess severity of LUTS in patients with symptomatic BPH using IPSS score before and after antibiotic therapy.

DETAILED DESCRIPTION:
This was a hospital-based prospective observational study.

All patients with symptomatic BPH attending the Urology Out-Patient Department (OPD) of the study site were enrolled. Informed and written consent was obtained from all participants. Demographic data were recorded, and detailed histories were taken regarding the duration and symptoms of BPH, including incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining, nocturia, and relevant past history. IPSS scoring was conducted. A thorough clinical examination, including general physical, systemic, and digital rectal examination, was performed. During the rectal examination, the prostate was checked for nodules, softness, induration, or tenderness. Urine culture and antibiotic sensitivity tests were conducted to assess the bacteriological profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic BPH.

Exclusion Criteria:

* Patients with indwelling catheters
* Recent antibiotic use
* Immunocompromised states (e.g., HIV, HCV)
* Uncontrolled diabetes mellitus (Hemoglobin A1c > 7%)
* Steroid therapy
* Those who declined to provide consent

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patient with Benign Prostate Hyperplasia
Study Population: All patients with symptomatic BPH attending the Urology Out-Patient Department (OPD) of the study site were enrolled. Informed and written consent was obtained from all participants. Demographic data were recorded, and detailed histories were taken. IPSS scoring was conducted. A thorough clinical examination, including general physical, systemic, and digital rectal examination, was performed. During the rectal examination, the prostate was checked for nodules, softness, induration, or tenderness. Urine culture and antibiotic sensitivity tests were conducted to assess the bacteriological profile. The patients was started on antibiotic therapy for a week based on antibiotic susceptibility testing.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Identification of common pathogens and Antibiotic susceptibility testing | 4 weeks
  Urine culture and antibiotic sensitivity tests were conducted to assess the bacteriological profile among symptomatic patients with BPH.

SECONDARY OUTCOMES:
Severity of LUTS in patients with symptomatic BPH | 4 weeks
  The study assess severity of LUTS in patients with symptomatic BPH using IPSS score before and after antibiotic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- BP Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) to be shared from this study will encompass demographic details (age, sex), clinical characteristics (severity and duration of lower urinary tract symptoms, baseline IPSS scores), microbiological findings (bacterial species isolated from urine cultures, antibiotic sensitivity patterns), treatment information (antibiotic regimen and duration), and clinical outcomes (post-treatment IPSS scores, follow-up urine culture results). This comprehensive dataset will facilitate in-depth analysis of the impact of antibiotic therapy on symptom relief and bacteriuria in patients with symptomatic Benign Prostatic Hyperplasia (BPH), thereby supporting future research and enhancing clinical management strategies.
Supporting Information: Study Protocol
Time Frame: Data will be made available after publication of manuscript in the journal.
Access Criteria: Researchers must provide a clear scientific rationale for requesting the data. Data will be shared upon reasonable request to the corresponding author. Requests must detail the intended use of the data and ensure it aligns with the ethical guidelines, ensuring patient confidentiality.